CLINICAL TRIAL: NCT06850779
Title: Effects of Radial Extracorporeal Shock Wave and Kinesio Taping Treatments on Quality of Life, Hand Function and Median Nerve Cross-Sectional Area Measured by Ultrasonography in Patients With Carpal Tunnel Syndrome: A Single-Blind Randomized Controlled Trial
Brief Title: Effects of Radial Extracorporeal Shock Wave and Kinesio Taping Treatments in Patients With Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Selda Çiftci, Medical doctor, Sisli Hamidiye Etfal Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 26.09.2023/4106
Record Dates: First submitted 2025-02-22; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Carpal Tunnel Syndrome (CTS)
Keywords: carpal tunnel syndrome; extracorporeal shock wave therapy; kinesio taping
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Extracorporeal Shockwave Therapy; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group 1 (Active Comparator): Those who received both extracorporeal shock wave therapy (ESWT) and kinesio taping (KB)
  Interventions: Other: Extracorporeal shock wave therapy (ESWT); Other: Kinesio taping (KT); Other: Exercise
- Group 2 (Active Comparator): Those who received ESWT
  Interventions: Other: Extracorporeal shock wave therapy (ESWT); Other: Exercise
- Group 3 (Active Comparator): Those who received KT
  Interventions: Other: Kinesio taping (KT); Other: Exercise
- Group 4 (Other): Those who received only exercise
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Extracorporeal shock wave therapy (ESWT) — Radial ESWT (Vibrolith OrthoⓇ) was applied to the wrist as 1000 pulses with a frequency of 5 Hz and a power of 1.5 bar. The treatment was applied once a week for a total of 3 sessions.
  Arms: Group 1; Group 2
Other: Kinesio taping (KT) — KT was prepared as 2 pieces of 2.5 cm I band and 1 piece of 5 cm I band. It was applied with a maximum of 50% tension (without tension on the ends) while the wrist was in 30 degrees of extension, forearm supination and elbow extension. The treatment was applied once a week for a total of 3 sessions.
  Arms: Group 1; Group 3
Other: Exercise — Median nerve gliding exercises were given to the 4th group during the follow-up period. The same exercises were given to the other groups.

SUMMARY:
Carpal Tunnel Syndrome (CTS) is a common upper extremity nerve compression syndrome that causes significant economic and social burden to affected individuals. Although the severity may vary among patients, symptoms such as night pain, transient numbness, tingling, constant pain, muscle weakness, and sleep disturbance may be observed. The treatment of CTS can be grouped as nonsurgical and surgical treatments. The aim of this study is to investigate the effects of treatment with sound waves and a healing method called extracorporeal shock wave therapy and a therapeutic flexible tape called kinesiology taping on pain, grip strength, quality of life, depression symptoms, hand functions, and ultrasonographic median nerve cross-sectional area in patients with CTS.

DETAILED DESCRIPTION:
Carpal tunnel syndrome is the most common nerve entrapment syndrome, typically affecting the dominant extremity. Symptoms often become more pronounced at night, and may include numbness, tingling, electric shock sensations, pain, and other related symptoms. Diagnosis can be made based on patient history, physical examination, electrodiagnostic tests, and ultrasonography. Treatment options include splinting, exercise therapy, physical therapy modalities, various injections, and surgical methods.

In our study, we compared the effects of extracorporeal shock wave therapy (ESWT) and kinesiology taping (KT) on carpal tunnel syndrome. The study involved four randomized groups: Group 1 received both ESWT and KT, Group 2 received only ESWT, Group 3 received only KT, and Group 4 received exercise therapy alone. Evaluations were conducted using the Visual Analog Scale, Boston Carpal Tunnel Questionnaire, Douleur Neuropathique 4 Questions, Nottingham Health Profile, grip strength measurements, and median nerve cross-sectional area via ultrasonography. Evaluations were performed three times: before treatment, at week 3, and at week 6.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate unilateral carpal tunnel syndrome confirmed by electroneuromyography (ENMG)
* Patients over 18 years of age
* Symptom duration of at least 3 months
* Those who have not received any medical treatment other than analgesics in the last 3 months

Exclusion Criteria:

* Bilateral Carpal Tunnel Syndrome (CTS)
* Severe CTS detected by ENMG
* Operated CTS
* Corticosteroid injection within the last 3 months
* History of peripheral nerve damage
* Secondary CTS causes (thyroid dysfunction, connective tissue diseases)
* Cervical disc herniation
* DeQuervain tenosynovitis, trigger finger, Dupuytren contracture
* Inflammatory disorder
* Bleeding disorder
* Pregnancy
* Malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Pain level before treatment, 3rd week and 6th week after treatment | From enrollment to the end of treatment at 3rd week and 6th week
  Pain level will be evaluated with the Visual Analog Scale. (minimum: 0, maximum: 100 mm)
Assessment of symptom severity and functionality | From enrollment to the end of treatment at 3rd week and 6th week
  The Boston Carpal Tunnel Syndrome Questionnaire (BCTQ) questionnaire was used to assess symptom severity and functionality. It includes 2 subgroups: Symptom Severity Scale (SSS) and Functional Status Scale (FSS). Symptom severity is assessed with 11 questions, and functional status is assessed with 8 questions. Each question is scored from low to high, 1 to 5. As the total score increases, deterioration increases.
Assessment of median nerve cross sectional area by ultrasonography | From enrollment to the end of treatment at 3rd week and 6th week
  The median nerve cross-sectional area was measured by tracing just proximal to the carpal tunnel entrance with the wrist resting on a table in a neutral position. The carpal tunnel entrance was identified by detecting the proximal side of the transverse carpal ligament. The distal radioulnar joint was also observed at this level.

SECONDARY OUTCOMES:
Assessment of grip strength and lateral pinch strength | From enrollment to the end of treatment at 3rd week and 6th week
  A hydraulic hand dynamometer was used to assess grip strength, and a hydraulic pinchmeter was used to assess lateral pinch strength. Measurements were made using the 2nd level resistance (3.75 cm) with the elbow at 90 degrees of flexion and the forearm and wrist in a neutral position. Patients were asked to squeeze with maximum force, measurements were made three times, and the average result was recorded in kilograms. For lateral pinch (LP), the pinchmeter was pressed with the distal middle of the thumb, and the lateral part of the second phalanx of the index finger was used to support the lower part.
Assessment of functionality | From enrollment to the end of treatment at 3rd week and 6th week
  Duruöz Hand Index was used for functional assessment. This questionnaire contains 18 questions on hand activities. It consists of five areas. There are eight questions on kitchen activities, two questions on dressing, two questions on personal hygiene, two questions on office work and four questions on other activities. The patient selects one of the answers for each question on a scale of one to five. The scores given for each question are added to obtain a total score ranging from 0 to 90. Higher scores indicate more severe hand disability.
Assessment of neuropathic pain | From enrollment to the end of treatment at 3rd week and 6th week
  Douleur Neuropathique 4 Questions was used to assessment of neuropathic pain. The DN4 questionnaire consists of 10 items. The first 7 items are related to pain characteristics and sensation, while the remaining 3 items are related to examination. For each item, a score of "1" is given if the answer is "yes" and a score of "0" if the answer is "no". If the total number of yes answers from the 10 items is calculated as 4 or more, the patient is defined as having neuropathic pain.
Assessment of quality of life | From enrollment to the end of treatment at 3rd week and 6th week
  The Nottingham Health Profile was used.As a general health status questionnaire, it provides a brief indication of a patient's perceived emotional, social and physical health and is designed for use in the general population. It is concerned with the individual's health status and includes energy levels, pain, emotional responses, sleep, social isolation and physical abilities. The energy levels domain consists of 3 items, pain 8 items, emotional responses 9 items, sleep and social isolation domains 5 items each and physical abilities domain 8 items. Each item requires a yes or no response. The patient's score is calculated out of a total of 600 points. The higher the score, the lower the quality of life.
Assessment of depression | From enrollment to the end of treatment at 3rd week and 6th week
  Beck Depression Inventory was used for depression assessment. It consists of 21 items with four precursors scored between 0 and 3. Patients are asked to mark the item that best suits their mood in the past week. As the score increases, it is thought that the depressive state is more severe. The total score is scored as 0-9 = Minimal, 10-16 = mild, 17-29 = moderate, 30-63 = severe.

CONTACTS AND LOCATIONS:
Overall Officials: Banu Kuran, Professor, MD, Study Director — Şişli Hamidiye Etfal Training and Research Hospital, Deparment of Physical Medicine and Rehabilitation
Locations (1):
- Şişli Hamidiye Etfal Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided